CLINICAL TRIAL: NCT01279590
Title: A Double-blind, Randomized, Placebo-controlled and Active-comparator-controlled Phase 2b Study to Evaluate Statin-associated Myalgia Incidence, Lipid Profile Effect, and Safety and Tolerability Associated With PPD10558 Versus Atorvastatin in Patients With Primary Hypercholesterolemia, Fredrickson IIa or IIb, Who Have Discontinued Two or More Prior Statin Therapies Due to Statin-associated Myalgia
Brief Title: Study of the Safety and Tolerability Associated With PPD10558 Versus Atorvastatin in Patients Previously Intolerant to Statins Due to Statin-associated Myalgia (SAM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Furiex Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPD10558-010
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Myalgia; Hypercholesterolemia; Hyperlipidemia
Keywords: Hyperlipidemia; Dyslipidemia; Metabolic diseases; Lipid metabolism disorders; Hyperlipoproteinemia Type IIa; Hyperlipoproteinemia Type IIb; Hypercholesterolemia, Autosomal Dominant; Hypercholesterolemia, Autosomal Dominant, Type B; Frederickson Type IIa; Frederickson Type IIb Hyperlipidemia
MeSH Terms: conditions — Myalgia; Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Metabolic Diseases; Lipid Metabolism Disorders; Hyperlipoproteinemia Type II | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PPD10558 (Experimental): Dosing will be forced-titrated as follows: 40 mg orally twice daily for 4 weeks and 80 mg orally twice daily for 8 weeks
  Interventions: Drug: PPD10558
- Atorvastatin (Active Comparator): Dosing will be forced titrated as 40 mg orally once daily for 4 weeks, and 80 mg orally once daily for 8 weeks
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Dosing will be 2 placebo capsules twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PPD10558 — PPD10558 40 mg capsule and matching placebo capsule twice a day for 4 weeks, then
  PPD10558 80 mg (two 40 mg capsules) twice a day for 8 weeks
  Arms: PPD10558
Drug: Atorvastatin — Atorvastatin 40 mg capsule and matching placebo capsule in the morning and 2 placebo capsules in the evening for 4 weeks, then
  Atorvastatin 80 mg (two 40 mg capsules) in the morning and 2 placebo capsules in the evening for 8 weeks
  Arms: Atorvastatin
Drug: Placebo — 2 placebo capsules twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the incidence of statin-associated myalgia (SAM) with treatment with PPD10558 versus atorvastatin in patients previously intolerant to statins.

To assess the safety and tolerability of PPD10558 compared to atorvastatin in patients previously intolerant to statins.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary hypercholesterolemia (heterozygous familial and nonfamilial) Fredrickson types IIa or IIb.
* history of statin-associated myalgia, as defined by being unable to tolerate two previous statins due to muscle pain, aches, weakness, or cramping that begins or increases during statin therapy and stops when statin therapy is discontinued. History of statin-associated myalgia will be captured on the historical questionnaire on statin-associated myalgia.
* LDL-C > 110 mg/dL and triglycerides < 500 mg/dL at Prescreening.
* prescreening hemoglobin value of ≥10 g/dL for females and ≥12 g/dL.
* patient agrees to stop all other antihyperlipidemic agents (including but not limited to niacin, probucol, ezetimibe, fibrates and derivatives, bile acid-sequestering agents, other 3-hydroxy-3-methylglutaryl-coenzyme A(HMG-CoA) reductase inhibitors, fish oils, flaxseed oil, and red yeast rice).
* patient agrees to stop all Coenzyme Q10 supplements.
* if taking other nonexcluded medications, patients must be on a stable dose for 4 weeks before screening.

Exclusion Criteria:

* history of chronic pain and currently experiences chronic pain unrelated to statins that requires chronic use of pain medications, has been diagnosed with fibromyalgia or has severe neuropathic pain.
* requires the chronic use of pain medications, including acetaminophen, non-steroidal anti-inflammatory medications, narcotics, and other analgesics.
* vitamin D insufficiency (current insufficiency is defined as Vitamin D3 < 20 ng/mL [50 nmol/L] measured at Prescreening.
* hypothyroidism or abnormal thyroid function test as confirmed by thyroid-stimulating hormone ≥ 5 mcIU/mL and free thyroxine (T4) < 0.7 ng/dL at Prescreening
* history of rhabdomyolysis (defined as evidence of organ damage with creatinine kinase(CK) > 10,000 IU/L).
* history of liver disease
* history of significant renal dysfunction as defined by serum creatinine clearance < 30 mL/min
* Nephrotic-range proteinuria.
* HbA1C >9% at Prescreening.
* CK levels >5 times the upper limit of normal at Prescreening.
* congestive heart failure, even with current therapy
* has had myocardial infarction, cardiac intervention, cerebrovascular accident/stroke or transient ischemic attack less than 6 months prior to prescreening.
* patient is pregnant (confirmed by laboratory testing) or breastfeeding.
* history of cancer (other than basal cell and/or squamous cell carcinoma of the skin and/or Stage I squamous cell carcinoma of the cervix) that has not been in full remission for at least 1 year before Screening.
* patient has positive test results for hepatitis B surface antigen (HBsAg), hepatitis C antibody, or human immunodeficiency virus types 1 or 2 at Prescreening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of stopping treatment with double-blinded study drug due to statin-associated myalgia. | Up to week 12
  Patients who withdraw from participating in the study prior to Week 12 and who also stop study drug due to SAM, or patients who become lost to follow up will be considered to have stopped treatment with double-blinded study drug.

SECONDARY OUTCOMES:
Change from Baseline in fasting lipid profile components (low density lipoprotein-cholesterol(LDL-C), high density lipoprotein-cholesterol(HDL-C), triglyceride(TG), total cholesterol(TC), Apolipoprotein B(ApoB), HDL-TG, LDL/HDL ratio and TC/HDL ratio) | Up to week 12
Change from baseline in muscle strength measurements (Sit-to-stand(STS) performance and hand grip strength by Jamar Hydraulic Hand Dynamometer) | Up to week 12
Frequency of pain rescue medication | Up to week 12
Change from Baseline in inflammatory markers (Tumor necrosis factor α (TNF-α), C-reactive protein (CRP), and lipoprotein-associated phospholipase A2 (Lp-PLA2)) | Up to week 12
Change in patients' functional health and well-being as measured by the Short Form-36v2 Health Survey (SF-36) | Up to week 12
Time to onset of statin -associated myalgia (SAM) | Up to week 12
Time to stopping treatment with study drug due to SAM | Up to week 12

CONTACTS AND LOCATIONS:
Locations (63):
- United States (63):
  - Furiex research site, Anniston, Alabama
  - Furiex research site, Phoenix, Arizona
  - Furiex research site, Huntington Park, California
  - Furiex research site, Long Beach, California
  - Furiex research site, Pismo Beach, California
  - Furiex research site, San Diego, California
  - Furiex research site, West Lake Village, California
  - Furiex research site, Colorado Springs, Colorado
  - Furiex research site, Golden, Colorado
  - Furiex research site, Hartford, Connecticut
  - Furiex research site, Boynton Beach, Florida
  - Furiex research site, Coral Gables, Florida
  - Furiex research site, Deerfield Beach, Florida
  - Furiex research site, Fort Lauderdale, Florida
  - Furiex research site, Gainesville, Florida
  - Furiex research site, Opa-locka, Florida
  - Furiex research site, Pembroke, Florida
  - Furiex research site, Sanford, Florida
  - Furiex research site, West Palm Beach, Florida
  - Furiex research site, Honolulu, Hawaii
  - Furiex Research site, Boise, Idaho
  - Furiex research site, Nampa, Idaho
  - Furiex research site, Chicago, Illinois
  - Furiex research site, Mission, Kansas
  - Furiex research site, Madisonville, Kentucky
  - Furiex research site, Covington, Louisiana
  - Furiex research site, Auburn, Maine
  - Furiex research site, Oxon Hill, Maryland
  - Furiex research site, Bay City, Michigan
  - Furiex research site, St Louis, Missouri
  - Furiex research site, Billings, Montana
  - Furiex research site, Butte, Montana
  - Furiex research site, Missoula, Montana
  - Furiex research site, Omaha, Nebraska
  - Furiex research site, Great Neck, New York
  - Furiex research site, Asheville, North Carolina
  - Furiex research site, Cary, North Carolina
  - Furiex research site, Charlotte, North Carolina
  - Furiex research site, Harrisburg, North Carolina
  - Furiex research site, Hickory, North Carolina
  - Furiex research site, High Point, North Carolina
  - Furiex research site, Raleigh, North Carolina
  - Furiex research site, Wilmington, North Carolina
  - Furiex research site, Carlisle, Ohio
  - Furiex research site, Cincinnati, Ohio
  - Furiex research site, Columbus, Ohio
  - Furiex research site, Kettering, Ohio
  - Furiex research site, Springfield, Ohio
  - Furiex research site, Altoona, Pennsylvania
  - Furiex research site, Johnstown, Pennsylvania
  - Furiex research site, Cumberland, Rhode Island
  - Furiex research site, East Providence, Rhode Island
  - Furiex research site, Anderson, South Carolina
  - Furiex research site, Greenville, South Carolina
  - Furiex research site, Greer, South Carolina
  - Furiex research site, Mt. Pleasant, South Carolina
  - Furiex research site, Pawleys Island, South Carolina
  - Furiex research site, Bristol, Tennessee
  - Furiex research site, Tomball, Texas
  - Furiex research site, Salt Lake City, Utah
  - Furiex research site, Norfolk, Virginia
  - Furiex research site, Richmond, Virginia
  - Furiex, Spokane, Washington